CLINICAL TRIAL: NCT03823950
Title: A Pilot Study of Granulocyte Colony-Stimulating Factor Starting at 24 Hours vs 72 Hours in Pediatric Oncology Patients
Brief Title: Starting Granulocyte Colony-Stimulating Factor at 1 Day vs 3 Days Following Chemotherapy in Pediatric Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0082
Record Dates: First submitted 2019-01-08; First posted 2019-01-31 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Granulocyte Colony-Stimulating Factor; Chemotherapy-induced Neutropenia; Chemotherapy-Induced Febrile Neutropenia; Pediatric Cancer
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Neoplasms | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Receive G-CSF 72 hours following chemotherapy (Experimental): Children will be enrolled during the first four rounds of chemotherapy. Upon enrollment, children will receive G-CSF at 24 hours following chemotherapy. G-CSF will be discontinued when absolute neutrophil count (ANC) has increased post nadir in accord with G-CSF administration guidelines. Parents and children will then complete questionnaires to determine rates of side effects and needle distress at the end of G-CSF during their next regular outpatient oncology clinic visit.
  Following children's next course of chemotherapy, G-CSF will be started 72 hours after completion of chemotherapy.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor
- Historical Controls (No Intervention): Four matched historical controls who received G-CSF at 24 hours following chemotherapy for each patient enrolled will be selected as each enrolled patient completes G-CSF therapy.

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor — Begin G-CSF 72 hours following chemotherapy
  Other Names: G-CSF
  Arms: Receive G-CSF 72 hours following chemotherapy

SUMMARY:
Chemotherapy places patients at an increased risk of infection. A medication called granulocyte colony-stimulating factor is given as a daily injection in order to help decrease the risk of infection. The purpose of this study is to determine the best time to begin granulocyte colony-stimulating factor while maintaining the same clinical benefits. The current study aims to fill these research gaps and address the general question: Can G-CSF safely be given 72 hours following the last day of chemotherapy without increasing the incidence of febrile neutropenia, the duration of neutropenia, or causing increased delays in the next course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oncology patients will be eligible to participate in this study if they meet the following inclusion criteria:

  1. are between the ages of birth and 21 years old
  2. is diagnosed with an oncologic disease
  3. is being treated at UMMC Children's Cancer Clinic
  4. will receive G-CSF as part of their standard or experimental oncology treatment protocol between January 1, 2019 and December 31, 2019. Oncology treatment protocols are typically derived from the Children's Oncology Group standard of care or patients can be enrolled on a Children's Oncology Group treatment study.
  5. is within first four courses of chemotherapy treatment

Exclusion Criteria:

* Patients will be excluded from the current study if:

  1. G-CSF was added to their oncology treatment protocol due to previous complications but for whom G-CSF was not part of their original treatment protocol.
  2. are being treated for relapsed disease
  3. has clinical evidence of bone marrow involvement

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital admissions for febrile neutropenia | From date of completion of course of chemotherapy until date of the initiation of next chemotherapy course, assessed up to 1 year
  Febrile neutropenia is defined as a temperature greater than or equal to 38 degrees Celsius and ANC less than or equal to 500

SECONDARY OUTCOMES:
Duration of neutropenia | From date of first recorded ANC following chemotherapy until date of first ANC that is greater than 500 following nadir, assessed up to 1 year
  The number of days between the first documented ANC less than or equal to 500 and the first documented ANC greater than 500 following nadir
Days delayed in beginning the next course of chemotherapy | Will be assessed weekly until the next course of chemotherapy is initiated, up to 1 year
  A delay in chemotherapy is defined when the initiation of the next course of chemotherapy is delayed due to neutropenia

OTHER OUTCOMES:
Needle distress | 2 days
  Distress Rating Tool: The DRS version for 2-, 3-, and 4-year-olds has three faces with different facial expressions for children to point to the one that best matches how they feel. The version for 5- and 6-year-olds has a visual analog scale presented as a thermometer with a happy face drawn next to the 0 and a sad face drawn next to the 10. The DRT version for youth 7 to 18 years defines distress as 'worry, anxiety, sadness, or fear,' on a scale from 0 (no distress) to 5 (moderate distress) to 10 (high distress). The adult DRS will be used for youth 19 to 21 years. Caregivers will rate their perception of their child's distress
Physical Side Effects | 1 week
  Memorial Symptom Assessment Scale: Physical and psychological symptoms; 8 items on 3-4 point scale (7-12 yrs) during past 2 days; 22 items on 4-5 point scale (10-14 yrs) during past week

CONTACTS AND LOCATIONS:
Overall Officials: Anderson B Collier, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Univeristy of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No